CLINICAL TRIAL: NCT01346709
Title: Prospective Evaluation of a RIsk Score for Postoperative Pulmonary COmPlications in Europe: Predicting Postoperative Pulmonary Complications in Europe: a 7-day Data Collection, Prospective, Observational Study
Brief Title: Prospective Evaluation of a RIsk Score for Postoperative Pulmonary COmPlications in Europe
Acronym: PERISCOPE
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: PERISCOPE
Record Dates: First submitted 2011-04-20; First posted 2011-05-03 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2015-10

CONDITIONS: Complication of Surgical Procedure; Acute Respiratory Failure, Adult; Postoperative Respiratory Complications; Pulmonary Failure; Surgical Complications From General Anesthesia
Keywords: Operative surgical procedures; Postoperative pulmonary complications (PPC); Epidemiological Study; ARISCAT score; Risk Score; Europe; PERISCOPE; observational study; Mild respiratory failure; Severe respiratory failure; acute lung injury (ALI); Acute respiratory distress syndrome (ARDS); Suspected pulmonary infection; Pulmonary infiltrate; Pleural effusion; Atelectasis; Pneumothorax; Bronchospasm; Aspiration Pneumonitis; Cardiopulmonary edema; Prospective Evaluation; nonobstetric in-hospital surgical procedure; general or regional anaesthesia; continued 7-day period recruitment
MeSH Terms: conditions — Respiratory Insufficiency; Acute Lung Injury; Respiratory Distress Syndrome; Pleural Effusion; Pulmonary Atelectasis; Pneumothorax; Bronchial Spasm; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In-patient Adult Non-obstetricSurgical: Consecutive patients admitted to participating centres undergoing surgery Non-obstetric in-hospital surgical procedure, elective or emergent, under general anaesthesia (alone or in combination with regional/neuraxial anaesthesia), neuraxial anaesthesia or plexus block (with and without sedation).
  All eligible patients undergoing surgery within the seven day study period will be recruited wherever possible.

SUMMARY:
Prospective Evaluation of a RIsk Score for postoperative pulmonary COmPlications in Europe (PERISCOPE) is a multi-centre, international observational study of a random-sample cohort of patients undergoing a nonobstetric in-hospital surgical procedure under general or regional anaesthesia during a continued 7-day period of recruitment.

DETAILED DESCRIPTION:
Prospective Evaluation of a RIsk Score for postoperative pulmonary COmPlications in Europe (PERISCOPE) is a multi-centre, international observational study of a random-sample cohort of patients undergoing a nonobstetric in-hospital surgical procedure under general or regional anaesthesia during a continued 7-day period of recruitment.

Participating centres throughout Europe will contribute routine clinical data describing all eligible patients who undergo surgery during a continuous week (7-days) at convenience of every department within a period of two months from May 1st to July 1st 2011. A questionnaire of around 50 items will be filled during the pre, intra and postoperative periods. The follow-up will end at discharge. The aim of the PERISCOPE study is to validate a simple score to predict postoperative pulmonary complications(PPCs). This score has recently been published in Anesthesiology and you can access linking to: http://journals.lww.com/anesthesiology/Fulltext/2010/12000/Prediction_of_Postoperative_Pulmonary.20.aspx

TIMEFRAME Participants will be followed for the duration of in-hospital stay, an expected average of maximum 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing a non-obstetric in-hospital surgical procedure, elective or emergent, under general anaesthesia (alone or in combination with regional/neuraxial anaesthesia), neuraxial anaesthesia or plexus block (with and without sedation).

Exclusion Criteria:

1. age <18 years
2. obstetric procedures or any procedure during pregnancy
3. regional anaesthesia alone, except to neuroaxial and plexus anaesthesia
4. procedures outside the operating room
5. procedures related to a previous postoperative complication
6. transplantation
7. patients with preoperatively intubated trachea
8. outpatient procedures, defined as those requiring less than one day's stay for a patient alive at discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patient adult non-obstetric surgery
Sampling Method: Probability Sample
Enrollment: 5450 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Canet, MD, Study Director — Hospital Universitari Germans Trias I Pujol, Barcelona, Spain; Sergi Sabaté, MD, PhD, Principal Investigator — Fundació Puigvert (IUNA), Barcelona, Spain; Olivier Langeron, MD, PhD, Principal Investigator — Groupe Hospitalier Pitie-Salpetriere; Marcelo Gama de Abreu, MD,PhD,DEAA, Principal Investigator — University Hospital Carl Gustav Carus Dresden University of Technology, Dresden, Germany; Lluís Gallart, MD, Principal Investigator — Parc de Salut Mar Anaesthesiology Research Group IMIM, Universitat Autònoma de Barcelona, Barcelona, Spain; Francisco Javier Belda, MD, Principal Investigator — Hospital Clínico Universitario de Valencia, Valencia, Spain; Paolo Pelosi, MD, PhD, Principal Investigator — University of Genoa, Genoa, Italy - San Martino Hospital, Genoa, Italy; Valentin Mazo, MD, Study Chair — Hospital Universitari Germans Trias I Pujol, Barcelona, Spain; Andreas Hoeft, MD, Principal Investigator — University Hospital, Bonn
Locations (63):
- University Hospital centre "Mother Theresa" Anesthesia & critical Care, Tirana, Albania
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- Bosnia and Herzegovina (2):
  - General Hospital "Prim.dr Abdulah Nakas" Departement of Anaesthesia and intensive care, Sarajevo
  - Heart Center, Sarajevo
- University Hospital Rijeka Anaesthesiology and Intensive care, Rijeka, Croatia
- Czechia (2):
  - Faculty Hospital Brno, department of Anaesthesiology and Intensive Care Medicine, Brno
  - Masaryks hospital Usti nad labem, Dept. of Anesthesia and intensive medicine, Ústí nad Labem
- Tartu University Hospital Clinic of Anaesthesiology and Intensive Care, Tartu, Estonia
- Hôpital Pitié-Salpêtrière, Anesthesiology and Critical Care, Paris, France
- Germany (4):
  - University Hospital Bonn, Anesthesiology, Bonn
  - Klinikum Darmstadt GmbH Anesthesiology, Intensive Care and pain medicin, Darmstadt
  - University Hospital Carl Gustav Carus, Dresden University of Technonology, Department of Anesthesiology and Intensive Care Therapy, Dresden
  - Universitätsmedizin Mainz, Departement of Anesthesiology, Mainz
- MISEK Kft., Anaesthesiology and Intensive Care Unit, Miskolc, Hungary
- Italy (8):
  - S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera S. Croce e Carle, Anesthesia, Cuneo
  - Ospedale San Martino, Dipartimento di scienze chirurgiche e diagnostiche integrate, Genoa
  - European Institute of Oncology,Anaesthesia and Intensive Care, Milan
  - University of Milano, Ospedale San Paolo Dpt Of Anaesthesia and Intensive Care, Milan
  - Azienda Ospedaliera Padova, Anesthesia and Intensive Care Clinic, Department of Pharmacology and Anesthesiology, Padua
  - Azienda USL n. 5 di Pisa Ospedale F. Lotti Anestesia e Rianimazione, Pontedera
  - University Of Insubria, Varese
- P Stradins Clinical University hospital, Departement of Anesthesiology, Riga, Latvia
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences, Clinic of Anaesthesiology, Kaunas
  - Vilnius University Hospital Santariskiu Clinics, Center of Anesthesiology, Intensive Care and Pain Treatment, Vilnius
- ZithaKlinik, Anaesthesiology and Intensive Care, Luxembourg, Luxembourg
- 10 Wojskowy Szpital Kliniczny z Polikliniką w Bydgoszczy, Anaesthesiology and Intensive Care, Bydgoszcz, Poland
- Portugal (4):
  - Hospitais da Universidade de Coimbra, EPE. Departement of Anesthesiology, Coimbra
  - Centro Hospitalar de Lisboa Ocidental, Serviço de Anestesia, Lisbon
  - Hospital Fernando Fonseca,Anesthesiology, Lisbon
  - Instituto Português de Oncologia, Departement of Anesthesiology, Porto
- Romania (3):
  - Emergency Institute of Cardiovascular Diseases Prof Dr C. C. Iliescu, Cardiac Anesthesia and Intensive Care, Bucharest
  - Emergency Clinical Hospital of Constanta, Department of Anaesthesiology and Intensive Care, Constanța
  - Emergency County Hospital Clinic of Anesthesia and Intensive Care, Intensive Care and Anesthesiology, Târgu Mureş
- Krasnoyarsk State Medical University,Anesthesiology and Intensive Care, Krasnoyarsk, Russia
- Spain (25):
  - Hospital General Universitario Alicante, Anaesthesiology, Alicante
  - Hospital Universitari Germans Trias i Pujol, Anaesthesiology, Badalona
  - Corporació Sanitària Parc Taulí, Anaesthesiology, Barcelona
  - Fundació Puigvert Anaesthesiology, Barcelona
  - Hospital Clinic, Anaesthesiology, Barcelona
  - Hospital Sant Pau, Anaesthesiology, Barcelona
  - Parc de Salut Mar, Anesthesiology, Barcelona
  - Vall d'Hebron University Hospital, Anaesthesiology, Barcelona
  - Hospital General de La Palma, Anestesiología y Reanimación, Breña Alta
  - Hospital de Denia,Anesthesia and Intensive Care, Denia
  - Hospital San Jorge, Anaesthesiology, Huesca
  - Hospital Arnau de Vilanova Departement of Anesthesiology, Lleida
  - Hospital Santa Maria, Departement of Anesthesiology, Lleida
  - Hospital 12 Octubre, Anaesthesiology, Madrid
  - Hospital del Tajo Anaesthesia and Reanimation, Madrid
  - Hospital Universitario de La Princesa, Anesthesiology, Madrid
  - Hospital Universitario de Móstoles, anestesiología y Reanimación, Madrid
  - Fundacio Althaia, Anaesthesiology, Manresa
  - Hospital Son Llatzer, Anaesthesiology, Palma de Mallorca
  - Clinica Universidad de Navarra, Anaesthesia, Pamplona
  - Hospital Universitario Marques De Valdecilla, Santander
  - Virgen del Rocio General Universitary Hospital;Anaesthesiology, Seville
  - Consorcio Hospital General Universitario, Anesthesiology, Critical Care and Pain Relief Unit, Valencia
  - Hospital Clínic Universitari de València, Anestesiología y Reanimación, Valencia
  - Hospital Universitario Rio Hortgea, Anaesthesia and Surgical Critical Care, Valladolid
- Ospedale Regionale di Lugano, Anestesia, Lugano, Switzerland
- Medical Faculty of Istanbul, Istanbul University, Anaesthesiology, Istanbul, Turkey (Türkiye)
- St.Katherine Hospital of Cardiology Anesthesiology & Pain Treatment, Odesa, Ukraine

REFERENCES:
- [Background] Canet J, Hardman J, Sabate S, Langeron O, Abreu MG, Gallart L, Belda J, Markstaller K, Pelosi P, Mazo V. PERISCOPE study: predicting post-operative pulmonary complications in Europe. Eur J Anaesthesiol. 2011 Jun;28(6):459-61. doi: 10.1097/EJA.0b013e328344be2d. No abstract available. PMID 21544025
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Result] Canet J, Sabate S, Mazo V, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P; PERISCOPE group. Development and validation of a score to predict postoperative respiratory failure in a multicentre European cohort: A prospective, observational study. Eur J Anaesthesiol. 2015 Jul;32(7):458-70. doi: 10.1097/EJA.0000000000000223. PMID 26020123
- [Result] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Derived] Russotto V, Sabate S, Canet J; PERISCOPE group; of the European Society of Anaesthesiology (ESA) Clinical Trial Network. Development of a prediction model for postoperative pneumonia: A multicentre prospective observational study. Eur J Anaesthesiol. 2019 Feb;36(2):93-104. doi: 10.1097/EJA.0000000000000921. PMID 30431500
- See also: The aim of the PERISCOPE study is to validate a simple score to predict postoperative pulmonary complications. This score has recently been published in Anesthesiology and you can access via this link — https://journals.lww.com/co-anesthesiology/Abstract/2019/06000/Prediction_of_postoperative_pulmonary.28.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 week chosen by each centre First Sub First Visit 4-Apr-11 Last data entered 25 Oct 2011
Period: Overall Study
Arm/Group | In-patient Adult Non-obstetricSurgical
Started | 5450
Completed | 5099
Not Completed | 351
Not completed — Protocol Violation | 35
Not completed — Lost to Follow-up | 31
Not completed — Missing data in candidate risk factor | 285

BASELINE CHARACTERISTICS:
Arm/Group | In-patient Adult Non-obstetricSurgical
Number analyzed (Participants) | 5099
Age, Customized [Number; unit: participants]
  <=50years | 1763
  51-80years | 2944
  >80years | 392
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age Median | 59.1 [44.9 to 70.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2493
  Male | 2606
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 26.2 [23.4 to 29.4]
Smoking status [Number; unit: participants]
  Never Smoker | 2674
  Former Smoker | 1245
  Current Smoker | 1180
Chronic obstructive pulmonary disease (COPD) [Number; unit: participants]
  COPD = yes | 517
  COPD = no | 4582
Functional Status [Number; unit: participants]
  Independant | 4561
  Partally/totally dependant | 538
Hypertension [Number; unit: participants]
  Hypertension = yes | 2191
  Hypertension = no | 2908
Heart Failure [Number; unit: participants]
  Heart Failure = yes | 800
  Heart Failure = no | 4299
Coronary artery disease [Number; unit: participants]
  Coronary artery disease = yes | 647
  Coronary artery disease = no | 4452
Cerebrovascular disease [Number; unit: participants]
  Cerebrovascular disease = yes | 654
  Cerebrovascular disease = no | 4445
Liver disease [Number; unit: participants]
  Liver disease = yes | 292
  Liver disease = no | 4807
Chronic kidney disease [Number; unit: participants]
  Chronic kidney disease = yes | 258
  Chronic kidney disease = no | 4841
Respiratory Infection in the last month [Number; unit: participants]
  Respiratory Infection in the last month = yes | 287
  Respiratory Infection in the last month = no | 4812
Preoperative SpO2 (Peripheral capillary oxygen saturation) [Median (Inter-Quartile Range); unit: Percentage] | 97 [96 to 99]
Anemia (<10g/dl) [Number; unit: participants]
  Anemia (<10g/dl) = yes | 223
  Anemia (<10g/dl) = no | 4876
Geografical Location of Centres [Number; unit: participants]
  Spain Centres | 2000
  Western Europe Centres | 1538
  Eastern Europe Centres | 1561
ASA physical status [Number; unit: participants] — a system for assessing the fitness of patients before surgery.
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  6. A declared brain-dead person whose organs are being removed for donor purposes.
  participants
    1 | 1115
    2 | 2604
    3 | 1280
    4 | 100
Anaesthesia [Number; unit: participants]
  General and combined | 3890
  Neuraxial/regional | 1209
Emergency Surgery [Number; unit: participants]
  Emergency Surgery = yes | 566
  Emergency Surgery = no | 4533
Surgical specialty [Number; unit: participants]
  Orthopedic | 998
  General and digestive | 1362
  Urology | 674
  Gynecology | 426
  Ear, nose, throat | 307
  Vascular | 201
  Breast | 153
  Cardiac | 161
  Thoracic | 142
  Neurosurgery | 320
  Other | 355
Surgical Incision [Number; unit: participants]
  Peripheral | 3695
  Upper abdominal | 1092
  Intrathoracic/cardiac | 312
Duration of Surgery (h) median [Median (Inter-Quartile Range); unit: hours] | 1.3 [0.8 to 2.3]

OUTCOME MEASURES:

1. Primary Outcome: The Main Outcome, Defined as a Postoperative Pulmonary Complications (PPC), Will be a Composite of the In-hospital Fatal or Non-fatal Postoperative Events.
Description: Will include:Mild respiratory failure;Severe respiratory failure;acute lung injury(ALI)/Acute respiratory distress syndrome(ARDS);Suspected pulmonary infection;Pulmonary infiltrate;Pleural effusion;Atelectasis;Pneumothorax;Bronchospasm;Aspiration Pneumonitis;Cardiopulmonary edema.Investigators will not modify centre usual patient management. Patients with PPCs will identify by consulting medical records and looking for events fulfilling PPCdefinition. Diagnosis date for every complication will be recorded.Participants will be followed during in-hospital stay up to 5 weeks.
Time Frame: Postoperative in-hospital stay up to 5 weeks
Population: PPC incidence, Percentage in Patients valid for external validation study
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | In-patient Adult Non-obstetricSurgical
Number analyzed (Participants) | 5099
Percentage of Participants | 7.92 [7.20 to 8.70]

2. Secondary Outcome: a) Postoperative Length of Stay
Description: Participants will be followed for the duration of in-hospital stay up to 90 days
Time Frame: Postoperative in-hospital stay up to 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | In-patient Adult Non-obstetricSurgical
Number analyzed (Participants) | 5099
days | 4 [2 to 7]

3. Secondary Outcome: b) In-hospital Mortality
Description: Participants will be followed for the duration of in-hospital stay up to 90 days
Time Frame: Postoperative in-hospital stay up to 90 days
Measure: Number; unit: percentage of Participants
Arm/Group | In-patient Adult Non-obstetricSurgical
Number analyzed (Participants) | 5099
percentage of Participants | 0.9

ADVERSE EVENTS:
Groups:
- Observational Study Section Not Applicable: observational study section not applicable
Arm/Group | Observational Study Section Not Applicable
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No